CLINICAL TRIAL: NCT04345445
Title: An Open-label, Randomized, Cross-over Interventional Study to Evaluate the Efficacy and Safety of Tocilizumab Versus Corticosteroids in Hospitalised COVID-19 Patients With High Risk of Progression
Brief Title: Study to Evaluate the Efficacy and Safety of Tocilizumab Versus Corticosteroids in Hospitalised COVID-19 Patients With High Risk of Progression
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Malaya (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: TVCS-COVID19
Record Dates: First submitted 2020-04-08; First posted 2020-04-14 (Actual); Last update posted 2020-04-14 (Actual); Status verified 2020-04

CONDITIONS: COVID-19
Keywords: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — tocilizumab; Methylprednisolone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tocilizumab (Experimental): Tocilizumab is given at 8 mg/kg (body weight) once and administered as an intravenous infusion within no less than 60 minutes.
  Interventions: Drug: Tocilizumab
- Methylprednisolone (Active Comparator): Reconstituted methylprednisolone is infused over 30 minutes and administered at a dose of 120mg/day for 3 days
  Interventions: Drug: Methylprednisolone

INTERVENTIONS:
Drug: Tocilizumab — IV infusion
  Arms: Tocilizumab
Drug: Methylprednisolone — IV infusion
  Arms: Methylprednisolone

SUMMARY:
This study aims to compare the efficacy and safety of Methylprednisolone versus Tocilizumab in improving clinical outcomes and reducing the need for ventilator support in COVID-19 patients with moderate COVID-19 disease at risk for complications of cytokine storm. Approximately 310 participants hospitalized with COVID-19 in UMMC, Hospital Sungai Buloh, Hospital Kuala Lumpur and Hospital Tuanku Jaafar will be enrolled into this study.

Eligible participants will be selected based on a set of clinical, laboratory and radiological parameters indicative of early stages of CRS and lung function decline prior to being randomized at a ratio of 1:1 to receive either Tocilizumab or Methylprednisolone. Participants will be monitored daily for clinical and laboratory parameters, and at 48 hours, switched to the alternate study arm should they manifest signs and symptoms indicative of decompensation.

ELIGIBILITY:
Inclusion Criteria:

1) Hospitalised symptomatic COVID-19 patients 2( Presence of clinical and radiological signs of progressive disease, AND laboratory evidence indicative of risk for cytokine storm complications.

All patients participating in this clinical trial must meet the following inclusion criteria:

1. Hospitalised symptomatic COVID-19 patients
2. Presence of clinical and radiological signs of progressive disease, AND laboratory evidence indicative of risk for cytokine storm complications:

   Clinical:

   Dyspnoea OR RR>20 breaths/min AND O2 sat <93% on RA OR increasing need for O2 supplementation to maintain O2 sat >95% on RA

   WITH

   Radiological:

   CXR or CT indicative of pneumonia OR worsening findings over time

   AND

   Laboratory:

   CRP levels >60 OR an increase of CRP >20 over 12 hours WITH an increasing ferritin level OR declining lymphocyte counts
3. Age > 18 years and able to give consent

Exclusion Criteria:

Patients will be excluded if any of the following conditions apply:

1. Known sensitivity/allergy to TCZ or other monoclonal antibodies
2. AST/ALT>5 times UNL, platelet counts <50,000 or neutrophil counts <500
3. Active TB
4. Pregnant
5. Receipt of mechanical ventilation
6. Has received other immunomodulatory drugs (including TCZ) in the past for the treatment of other conditions
7. Individuals, in the opinion of the investigator, where progression to death is imminent and inevitable in the next 24 hours irrespective of treatment provision or who have signed a DNR.
8. Participating in other clinical trials (subject to approval)
9. Any serious medical condition or abnormal clinical laboratory tests which in the judgement of the investigator may compromise patient safety should he/she participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 310 (Estimated)
Dates: Start 2020-04-15 (Estimated); Primary Completion 2020-10-31 (Estimated); Study Completion 2020-10-31 (Estimated)

PRIMARY OUTCOMES:
The proportion of patients requiring mechanical ventilation | Through study completion, and average of 6 months
Mean days of ventilation | Through study completion, and average of 6 months

SECONDARY OUTCOMES:
The proportion of patients requiring ICU admission | Through study completion, and average of 6 months
Overall 28-day survival | 28 day from baseline
Change in symptom severity assessed by the World Health Organization (WHO) Coronavirus Disease 2019 (COVID19) ordinal scale measured daily up to 7 days from baseline | 7 days from baseline
Duration of hospital and ICU stay | Through study completion, and average of 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- University Malaya Medical Centre, Kuala Lumpur, Malaysia

IPD SHARING:
Plan to Share IPD: Undecided